CLINICAL TRIAL: NCT02915705
Title: A Randomized, Open-Label, Phase 3 Study to Assess the Efficacy and Safety of KRN23 Versus Oral Phosphate and Active Vitamin D Treatment in Pediatric Patients With X Linked Hypophosphatemia (XLH)
Brief Title: Efficacy and Safety of Burosumab Versus Oral Phosphate and Active Vitamin D Treatment in Pediatric Patients With XLH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UX023-CL301
Expanded Access: NCT03775187 (Available)
Record Dates: First submitted 2016-05-23; First posted 2016-09-27 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: X-Linked Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Burosumab (Experimental): Burosumab 0.8 mg/kg starting dose, administered Q2W by SC injection during the Treatment Period (up to Week 64). During the Treatment Extension Period (Week 64 to Week 140), participants continued to receive a starting dose of SC burosumab 0.8 mg/kg Q2W. Participants in Japan and Korea did not enter the Treatment Extension Period.
  Interventions: Biological: burosumab
- Active Control (Active Comparator): Multiple daily doses of oral phosphate and one or more daily doses of active vitamin D therapy, titrated and individualized by the investigator based on published recommendations during the Treatment Period (up to Week 64). During the Treatment Extension Period (Week 64 to Week 140), participants crossed over to receive a starting dose of SC burosumab 0.8 mg/kg Q2W. Participants in Japan and Korea did not enter the Treatment Extension Period.
  Interventions: Biological: burosumab; Drug: Oral Phosphate Supplement; Drug: active vitamin D

INTERVENTIONS:
Biological: burosumab — solution for subcutaneous (SC) injection
  Other Names: KRN23; Crysvita ®; UX023
Drug: Oral Phosphate Supplement — oral tablet; oral solution; oral powder
  Arms: Active Control
Drug: active vitamin D — tablet, oral solution
  Arms: Active Control

SUMMARY:
The primary objective of this study is to evaluate the effect of KRN23 (burosumab) therapy in improving rickets in children with XLH compared with active control (oral phosphate/active vitamin D).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 1 to ≤12 years with radiographic evidence of rickets as determined by central readers
2. Phosphate-regulating endopeptidase homolog, X-linked (PHEX) mutation or variant of uncertain significance in either the patient or in a directly related family member with appropriate X-linked inheritance
3. Biochemical findings associated with XLH: serum phosphorus <3.0 mg/dL (<0.97 mmol/L)
4. Serum creatinine below the age-adjusted upper limit of normal
5. Serum 25(OH)D above the lower limit of normal (≥16 ng/mL) at the Screening Visit
6. Have received both oral phosphate and active vitamin D therapy for ≥ 12 consecutive months (for children ≥3 years of age) or ≥ 6 consecutive months (for children <3 years of age) 7 days prior to the Randomization Visit
7. Willing to provide access to prior medical records for the collection of historical growth and radiographic data and disease history
8. Provide written or verbal assent (as appropriate for the subject and region) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
9. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments
10. Females who have reached menarche must have a negative pregnancy test at Screening and undergo additional pregnancy testing during the study. Female subjects of childbearing potential must be willing to use a highly effective method of contraception for the duration of the study plus 12 weeks after stopping the study drug. Sexually active male subjects with female partners of childbearing potential must consent to use a condom with spermicide or a highly effective method of contraception for the duration of the study plus 12 weeks after stopping the study drug

Exclusion Criteria:

1. Tanner stage 4 or higher in any of the following: genitals, breast, or pubic hair, based on physical examination
2. Height percentile > 50th based on country-specific norms
3. Use of aluminum hydroxide antacids (eg, Maalox® and Mylanta®), systemic corticosteroids, acetazolamide, and thiazides within 7 days prior to the Screening Visit
4. Current or prior use of leuprorelin (eg, Lupron®, Viadur®, Eligard®), triptorelin (TRELSTAR®), goserelin (Zoladex®), or other drugs known to delay puberty
5. Use of growth hormone therapy within 12 months before the Screening Visit
6. Presence of nephrocalcinosis on renal ultrasound grade 4
7. Planned orthopedic surgery, including osteotomy or implantation or removal of staples, 8 plates, or any other hardware, within the first 40 weeks of the study
8. Hypocalcemia or hypercalcemia, defined as serum calcium levels outside the age-adjusted normal limits
9. Evidence of hyperparathyroidism (parathyroid hormone [PTH] levels 2.5X upper limit of normal [ULN])
10. Use of medication to suppress PTH (eg, cinacalcet, calcimimetics) within 2 months prior to the Screening Visit
11. Presence or history of any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study.
12. Presence of a concurrent disease or condition that would interfere with study participation or affect safety
13. History of recurrent infection or predisposition to infection, or of known immunodeficiency
14. Use of a therapeutic monoclonal antibody within 90 days prior to the Screening Visit or history of allergic or anaphylactic reactions to any monoclonal antibody
15. Presence or history of any hypersensitivity to KRN23 excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects
16. Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments. OR, in Japan, use of any investigational product or investigational medical device within 4 months prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (16):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF, San Francisco, California
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Shriners Hospital For Children, St Louis, Missouri
  - Vanderbilt Children's Hospital, Nashville, Tennessee
- The Children's Hospital at Westmead, Westmead, New South Wales, Australia
- Canada (3):
  - Children's Hospital of Eastern Ontario (CHEO) Research Institute, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Shriners Hospital for Children - Canada, Montreal, Quebec
- Japan (3):
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Okayama Saiseikai General Hospital, Okayama
  - Japan Community Healthcare Organization Osaka Hospital, Osaka
- Seoul National University Hospital, Seoul, South Korea
- Karolinska Institutet and University Hospital, Stockholm, Sweden
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Royal Manchester Children's Hospital - University of Manchester, Manchester

REFERENCES:
- [Derived] Imel EA, Glorieux FH, Whyte MP, Portale AA, Munns CF, Nilsson O, Simmons JH, Padidela R, Namba N, Cheong HI, Pitukcheewanont P, Sochett E, Hogler W, Muroya K, Tanaka H, Gottesman GS, Biggin A, Perwad F, Chen A, Roberts MS, Ward LM. Burosumab vs Phosphate/Active Vitamin D in Pediatric X-Linked Hypophosphatemia: A Subgroup Analysis by Dose Level. J Clin Endocrinol Metab. 2023 Oct 18;108(11):2990-2998. doi: 10.1210/clinem/dgad230. PMID 37084401
- [Derived] Ward LM, Glorieux FH, Whyte MP, Munns CF, Portale AA, Hogler W, Simmons JH, Gottesman GS, Padidela R, Namba N, Cheong HI, Nilsson O, Mao M, Chen A, Skrinar A, Roberts MS, Imel EA. Effect of Burosumab Compared With Conventional Therapy on Younger vs Older Children With X-linked Hypophosphatemia. J Clin Endocrinol Metab. 2022 Jul 14;107(8):e3241-e3253. doi: 10.1210/clinem/dgac296. PMID 35533340
- [Derived] Padidela R, Whyte MP, Glorieux FH, Munns CF, Ward LM, Nilsson O, Portale AA, Simmons JH, Namba N, Cheong HI, Pitukcheewanont P, Sochett E, Hogler W, Muroya K, Tanaka H, Gottesman GS, Biggin A, Perwad F, Williams A, Nixon A, Sun W, Chen A, Skrinar A, Imel EA. Patient-Reported Outcomes from a Randomized, Active-Controlled, Open-Label, Phase 3 Trial of Burosumab Versus Conventional Therapy in Children with X-Linked Hypophosphatemia. Calcif Tissue Int. 2021 May;108(5):622-633. doi: 10.1007/s00223-020-00797-x. Epub 2021 Jan 23. PMID 33484279
- [Derived] Mao M, Carpenter TO, Whyte MP, Skrinar A, Chen CY, San Martin J, Rogol AD. Growth Curves for Children with X-linked Hypophosphatemia. J Clin Endocrinol Metab. 2020 Oct 1;105(10):3243-9. doi: 10.1210/clinem/dgaa495. PMID 32721016
- [Derived] Imel EA, Glorieux FH, Whyte MP, Munns CF, Ward LM, Nilsson O, Simmons JH, Padidela R, Namba N, Cheong HI, Pitukcheewanont P, Sochett E, Hogler W, Muroya K, Tanaka H, Gottesman GS, Biggin A, Perwad F, Mao M, Chen CY, Skrinar A, San Martin J, Portale AA. Burosumab versus conventional therapy in children with X-linked hypophosphataemia: a randomised, active-controlled, open-label, phase 3 trial. Lancet. 2019 Jun 15;393(10189):2416-2427. doi: 10.1016/S0140-6736(19)30654-3. Epub 2019 May 16. PMID 31104833

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants discontinued oral phosphate and active vitamin D therapy for 7 days prior to randomization. Participants were then randomized 1:1 to receive either open label burosumab administered by subcutaneous (SC) injection every 2 weeks (Q2W) or phosphate and active vitamin D therapy administered orally daily for a total of 64 weeks.
Period: Treatment Period
Arm/Group | Active Control | Burosumab
Started | 32 | 29
Completed Week 40 | 32 | 29
Completed Week 64 | 32 | 29
Completed | 32 | 29
Not Completed | 0 | 0
Period: Long Term Extension Period
Arm/Group | Active Control | Burosumab
Started | 26 (6 participants did not enter the extension period) | 25 (4 participants did not enter the extension period)
Completed | 26 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Control | Burosumab | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — age at first dose
  years | 6.50 (3.250) | 6.01 (3.408) | 6.27 (3.307)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 2 | 8
  White | 25 | 25 | 50
  Other (Not Specified) | 1 | 2 | 3
Rickets Severity Score (RSS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The RSS system is a 10-point radiographic scoring method. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees (the total score is the sum of the wrist and knee score). Higher scores indicate greater rickets severity.
  score on a scale | 3.19 (1.141) | 3.17 (0.975) | 3.18 (1.057)
Height-For-Age Z-Score [Mean (Standard Deviation); unit: Z score] — Recumbent length/Standing height z scores are measures of height adjusted for a child's age and sex. The Z-score indicates the number of standard deviations away from a reference population (from the Centers for Disease Control [CDC] growth charts) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome. Population: 1 participant in the burosumab group did not have a baseline measurement
  Z score
    number analyzed (Participants) | 32 | 28 | 60
    (all) | -2.05 (0.868) | -2.32 (1.167) | -2.17 (1.018)
Growth Velocity Z Score From Pre-Treatment [Mean (Standard Deviation); unit: Z score] — The Z score indicates the number of standard deviations away from a reference population (from Tanner's standard) in the same age range and with the same sex. The baseline growth velocity was calculated for participants who had data available from within 1.5 years prior to baseline. Children with a mid-point age under 2.25 years were excluded, because younger ages are not available in Tanner's standard. A Z score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a better outcome. Population: participants with a baseline measurement
  Z score
    number analyzed (Participants) | 22 | 22 | 44
    (all) | -2.14 (5.571) | -1.37 (1.334) | -1.75 (4.022)
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] | 2.30 (0.257) | 2.42 (0.244) | 2.36 (0.256)
Serum 1,25(OH)D [Mean (Standard Deviation); unit: pg/mL] — Population: participants with a baseline measurement
  pg/mL
    number analyzed (Participants) | 30 | 28 | 58
    (all) | 40.18 (14.886) | 46.00 (20.060) | 42.99 (17.663)
Ratio of Renal Tubular Maximum Reabsorption Rate of Phosphate to Glomerular Filtration Rate(TmP/GFR) [Mean (Standard Deviation); unit: mg/dL] — Data for urinary phosphorus and tubular reabsorption of phosphate (TRP) were used in the calculation of TmP/GFR. Population: participants with a baseline measurement
  mg/dL
    number analyzed (Participants) | 30 | 24 | 54
    (all) | 2.008 (0.3300) | 2.193 (0.3733) | 2.091 (0.3587)
Serum Alkaline Phosphatase (ALP) Concentration [Mean (Standard Deviation); unit: U/L] | 523.44 (154.419) | 510.76 (124.903) | 517.4 (140.15)
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Pain Interference Domain [Mean (Standard Deviation); unit: T-score] — The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013), (NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Pain Interference Domain, decreases indicate less pain. Population: participants with a baseline assessment
  T-score
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 49.9 (12.05) | 53.1 (10.95) | 51.3 (11.54)
PROMIS Physical Function Mobility Domain [Mean (Standard Deviation); unit: T-score] — The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013), (NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Physical Function Mobility Domain, increases indicate greater mobility. Population: participants with a baseline assessment
  T-score
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 45.5 (9.86) | 45.2 (9.05) | 45.3 (9.39)
PROMIS Fatigue Domain [Mean (Standard Deviation); unit: T-score] — The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013), (NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Fatigue Domain, decreases indicate less fatigue. Population: participants with a baseline assessment
  T-score
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 47.0 (13.70) | 48.8 (9.60) | 47.8 (11.98)
Faces Pain Scale-Revised (FPS-R) [Mean (Standard Deviation); unit: score on a scale] — The FPS-R is a dimensionless 10 point Likert scale used to assess self-reported pain intensity on a scale from 0 (no pain) to 10 (most pain you can imagine). Greater pain scores are indicative of more severe pain. Population: participants with a baseline assessment
  score on a scale
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 0.7 (1.17) | 0.4 (1.12) | 0.6 (1.14)
Six Minute Walk Test (6MWT) Total Distance [Mean (Standard Deviation); unit: meters] — The total distance walked (meters) in a 6-minute period was measured, and the percent predicted distance based on normative data for age and gender was estimated. Population: participants with a baseline measurement
  meters
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 450.50 (106.432) | 365.93 (118.083) | 414.26 (117.790)
Percent of Predicted Normal in the 6MWT Total Distance [Mean (Standard Deviation); unit: perecent of predicted meters] — The total distance walked (meters) in a 6-minute period was measured, and the percent predicted distance based on normative data for age and gender was estimated. Population: participants with a baseline measurement
  perecent of predicted meters
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 76.20 (14.838) | 62.13 (18.629) | 70.17 (17.771)

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Global Impression of Change (RGI-C) Global Score at Week 40
Description: Changes in the severity of rickets and bowing were assessed using a disease specific qualitative RGI-C scoring system. The RGI-C is a 7-point ordinal scale with possible values: +3 = very much better (complete or near complete healing of rickets), +2 = much better (substantial healing of rickets), +1 = minimally better (i.e., minimal healing of rickets), 0 = unchanged, -1 = minimally worse (minimal worsening of rickets), -2 = much worse (moderate worsening of rickets), -3 = very much worse (severe worsening of rickets).
Time Frame: Week 40
Population: Full Analysis Set: all randomized participants who received at least one dose of assigned medication and had at least one post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
score on a scale | 0.77 (0.107) | 1.92 (0.110)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Least squares (LS) mean, standard error (SE), confidence interval (CI), and 2-sided p value per ANCOVA model, which included RGI-C as the dependent variable, treatment group and baseline age stratification factor as independent variables and baseline RSS score as a continuous covariate; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = 1.14, 95% CI 2-sided [0.83 to 1.45]

2. Secondary Outcome: Percentage of Participants With a Mean RGI-C Global Score ≥ +2.0 (Responders) at Week 40
Description: RGI-C responders are defined as participants with a mean RGI-C global score >= +2.0. The RGI-C is a 7-point ordinal scale with possible values: +3 = very much better (complete or near complete healing of rickets), +2 = much better (substantial healing of rickets), +1 = minimally better (i.e., minimal healing of rickets), 0 = unchanged, -1 = minimally worse (minimal worsening of rickets), -2 = much worse (moderate worsening of rickets), -3 = very much worse (severe worsening of rickets).
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
percentage of participants | 6.3 | 72.4
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Test type: Superiority; p < 0.0001, Regression, Logistic — Odds ratio, CI, and 2-sided p-value were per logistic regression model, which included treatment group and baseline age stratification factor as independent variables and baseline RSS score as a continuous covariate; Odds Ratio (OR) = 39.1, 95% CI 2-sided [7.2 to 211.7]

3. Secondary Outcome: Percentage of Participants With a Mean RGI-C Global Score ≥ +2.0 (Responders) at Week 64
Description: as for outcome 2
Time Frame: Week 64
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
percentage of participants | 18.8 | 86.2
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Test type: Superiority; p = 0.0002, generalized linear mixed model — Odds ratio, CI, and 2-sided p-value were per generalized linear mixed model, which includes treatment, visit, treatment by visit interaction and baseline age stratification factor as factors, baseline RSS total score as a continuous covariate; Odds Ratio (OR) = 34.1, 95% CI 2-sided [5.6 to 206.3]

4. Secondary Outcome: RGI-C Global Score at Week 64
Description: as for outcome 1
Time Frame: Week 64
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
score on a scale | 1.03 (0.136) | 2.06 (0.072)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Per generalized estimating equation (GEE) model, which included RGI-C as the dependent variable, treatment, visit, treatment by visit interaction and baseline age stratification factor as factors, baseline RSS score as a continuous covariate, with exchangeable covariate structure; Test type: Superiority; p < 0.0001, GEE model; difference in LS means = 1.02, 95% CI 2-sided [0.72 to 1.33]

5. Secondary Outcome: Change From Baseline in RSS Total Score at Week 40
Description: The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, lucency, separation, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees (the total score is the sum of the wrist and knee score). Higher scores indicate greater rickets severity.
Time Frame: Baseline, Week 40
Population: Full Analysis Set: all randomized participants who received at least one dose of assigned medication and had at least one post-baseline RSS Total Score assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 28
score on a scale | -0.71 (0.138) | -2.04 (0.145)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Test type: Superiority; p < 0.0001, ANCOVA — LS mean, SE, CI, and 2-sided p value per ANCOVA model, which included treatment group and baseline age stratification factor as independent variables and baseline RSS score as a continuous covariate; LS Mean Difference = -1.34, 95% CI 2-sided [-1.74 to -0.94]

6. Secondary Outcome: Change From Baseline in RSS Total Score at Week 64
Description: The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees. Higher scores indicate greater rickets severity.
Time Frame: Baseline, Week 64
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
score on a scale | -1.01 (0.151) | -2.23 (0.117)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Test type: Superiority; p < 0.0001, GEE model — LS mean, SE, CI, and 2-sided p value per GEE model, which included treatment, visit, treatment by visit interaction and baseline age stratification factor as factors, baseline RSS score as a continuous covariate; difference in LS means = -1.21, 95% CI 2-sided [-1.59 to -0.83]

7. Secondary Outcome: RGI-C Long Leg Score at Week 40
Description: Changes in the severity of lower extremity skeletal abnormalities, including genu varum and genu valgus, were assessed using a disease specific qualitative RGI-C scoring system. The RGI-C is a 7-point ordinal scale with possible values: +3 = very much better (complete or near complete healing), +2 = much better (substantial healing), +1 = minimally better (i.e., minimal healing), 0 = unchanged, -1 = minimally worse (minimal worsening), -2 = much worse (moderate worsening), -3 = very much worse (severe worsening).
Time Frame: Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
score on a scale | 0.22 (0.080) | 0.62 (0.153)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Test type: Superiority; p = 0.0162, GEE model — LS mean, SE, CI, and 2-sided p value per GEE model, which included treatment, visit, treatment by visit interaction, and baseline age stratification factor as factors; and baseline RSS score as a continuous covariate; LS Mean Difference = 0.40, 95% CI 2-sided [0.07 to 0.72]

8. Secondary Outcome: RGI-C Long Leg Score at Week 64
Description: as for outcome 7
Time Frame: Week 64
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
score on a scale | 0.29 (0.119) | 1.25 (0.170)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 7, analysis 1]; difference in LS means = 0.97, 95% CI 2-sided [0.57 to 1.37]

9. Secondary Outcome: Change From Baseline in Height-For-Age Z-Scores to Week 40
Description: Recumbent length/Standing height z scores are measures of height adjusted for a child's age and sex. The Z-score indicates the number of standard deviations away from a reference population (from the Centers for Disease Control [CDC] growth charts) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
Time Frame: Baseline, Week 40
Population: Full Analysis Set: all randomized participants who received at least one dose of assigned medication and had at least one post-baseline assessment. Participants with an assessment at Week 40.
Measure: Least Squares Mean (Standard Error); unit: Z score
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 28
Z score | 0.03 (0.031) | 0.16 (0.052)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; LS mean, SE, CI, and 2-sided p value per GEE model, which included change from baseline for recumbent length/standing height Z score as the dependent variable, treatment group, visit, interaction between treatment group by visit and baseline RSS stratification as factors, age and baseline recumbent length/standing height Z score as continuous covariates, with exchangeable covariance structure; Test type: Superiority; p = 0.0408, GEE model; LS Mean Difference = 0.12, 95% CI 2-sided [0.01 to 0.24]

10. Secondary Outcome: Change From Baseline in Height-For-Age Z-Scores to Week 64
Description: Recumbent length/Standing height z scores are measures of height adjusted for a child's age and sex. The Z-score indicates the number of standard deviations away from a reference population (from the CDC growth charts) in the same age range and with the same sex. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
Time Frame: Baseline, Week 64
Population: Full Analysis Set: all randomized participants who received at least one dose of assigned medication and had at least one post-baseline assessment. Participants with an assessment at Week 64.
Measure: Least Squares Mean (Standard Error); unit: Z score
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 28
Z score | 0.02 (0.035) | 0.17 (0.066)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0490, GEE model; difference in LS means = 0.14, 95% CI 2-sided [0.00 to 0.29]

11. Secondary Outcome: Change in Growth Velocity Z Score From Baseline to Week 40
Description: A growth velocity Z score was calculated based on Tanner's standard. The Z score indicates the number of standard deviations away from a reference population (from Tanner's standard) in the same age range and with the same sex. The baseline growth velocity was calculated for participants who had data available from within 1.5 years prior to baseline. The Week 64 growth velocity was calculated using data between baseline and Week 64. The mid-point of the age interval was used to locate the closest reference age provided by Tanner's Standard. Children with a mid-point age under 2.25 years were excluded, because younger ages are not available in Tanner's standard. To smoothly transition from recumbent length to standing height, 0·8 cm was subtracted from recumbent length before pooling with standing height. A Z score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a better outcome.
Time Frame: Baseline, Week 40
Population: Full Analysis Set: all randomized participants who received at least one dose of assigned medication and had at least one post-baseline assessment. Participants with Baseline growth velocity.
Measure: Least Squares Mean (Standard Error); unit: Z score
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 22 | 22
Z score | 0.73 (0.339) | 1.76 (0.337)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; LS mean, SE, CI, and 2-sided p value per ANCOVA model, which included change from baseline for growth velocity Z score as the dependent variable, treatment group and baseline RSS total score stratification as factors, baseline Z score and age as continuous covariates; Test type: Superiority; p = 0.0386, ANCOVA; difference in LS means = 1.02, 95% CI 2-sided [0.06 to 1.99]

12. Secondary Outcome: Change in Growth Velocity Z Score From Baseline to Week 64
Description: as for outcome 11
Time Frame: Baseline, Week 64
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Z score
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 22 | 22
Z score | 0.41 (0.265) | 1.53 (0.264)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0047, ANCOVA; difference in LS means = 1.12, 95% CI 2-sided [0.37 to 1.88]

13. Secondary Outcome: Change From Baseline Over Time in Serum Phosphorus Concentration, up to Week 64
Description: The GEE model includes change from baseline for serum phosphorous measurement as the dependent variable, treatment group, visit, interaction between treatment group by visit, baseline age and baseline RSS stratification as factors, baseline phosphorous measure as a covariate, with exchangeable covariance structure. The GEE model included data up to Week 64.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16, 24, 32, 33, 40, 52, 64
Population: Pharmacodynamic (PD) Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data. Participants with data at given time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
mg/dL
  Week 1: number analyzed (Participants) | 31 | 28
  Week 1 | 0.22 (0.072) | 1.26 (0.094)
  Week 2: number analyzed (Participants) | 0 | 26
  Week 2 |  | 1.14 (0.098)
  Week 4 | 0.18 (0.061) | 1.21 (0.102)
  Week 8 | 0.21 (0.064) | 0.99 (0.074)
  Week 12: number analyzed (Participants) | 0 | 26
  Week 12 |  | 1.01 (0.072)
  Week 16: number analyzed (Participants) | 29 | 29
  Week 16 | 0.24 (0.063) | 0.87 (0.072)
  Week 24 | 0.27 (0.073) | 0.78 (0.077)
  Week 32 | 0.23 (0.063) | 0.93 (0.073)
  Week 33: number analyzed (Participants) | 0 | 27
  Week 33 |  | 1.23 (0.106)
  Week 40 | 0.20 (0.062) | 0.92 (0.080)
  Week 52 | 0.30 (0.082) | 0.91 (0.075)
  Week 64 | 0.21 (0.062) | 0.91 (0.078)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Week 1; Test type: Superiority; p < 0.0001, GEE model; difference = 1.04, 95% CI 2-sided [0.81 to 1.27] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 2: Comparison: Active Control vs Burosumab; Week 4; Test type: Superiority; p < 0.0001, GEE model; difference = 1.03, 95% CI 2-sided [0.79 to 1.27] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 3: Comparison: Active Control vs Burosumab; Week 8; Test type: Superiority; p < 0.0001, GEE model; difference = 0.78, 95% CI 2-sided [0.58 to 0.97] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 4: Comparison: Active Control vs Burosumab; Week 16; Test type: Superiority; p < 0.0001, GEE model; difference = 0.63, 95% CI 2-sided [0.44 to 0.81] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 5: Comparison: Active Control vs Burosumab; Week 24; Test type: Superiority; p < 0.0001, GEE model; difference = 0.51, 95% CI 2-sided [0.30 to 0.72] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 6: Comparison: Active Control vs Burosumab; Week 32; Test type: Superiority; p < 0.0001, GEE model; difference = 0.70, 95% CI 2-sided [0.51 to 0.89]
Statistical Analysis 7: Comparison: Active Control vs Burosumab; Week 40; Test type: Superiority; p < 0.0001, GEE model; difference = 0.71, 95% CI 2-sided [0.51 to 0.91] — Difference (burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 8: Comparison: Active Control vs Burosumab; Week 52; Test type: Superiority; p < 0.0001, GEE model; difference = 0.61, 95% CI 2-sided [0.39 to 0.82]
Statistical Analysis 9: Comparison: Active Control vs Burosumab; Week 64; Test type: Superiority; p < 0.0001, GEE model; difference = 0.69, 95% CI 2-sided [0.49 to 0.90]

14. Secondary Outcome: Change From Baseline Over Time in Serum Phosphorus Concentration, Weeks 66-112
Time Frame: Baseline, Weeks 66, 68, 76, 88, 100, 112
Population: PD Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 26 | 22
mg/dL
  Week 66: number analyzed (Participants) | 26 | 0
  Week 66 | 0.05 (0.235) |
  Week 68: number analyzed (Participants) | 26 | 1
  Week 68 | 1.17 (0.472) | 1.10 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 22 | 22
  Week 76 | 0.90 (0.324) | 0.92 (0.324)
  Week 88: number analyzed (Participants) | 16 | 11
  Week 88 | 0.98 (0.433) | 1.00 (0.576)
  Week 100: number analyzed (Participants) | 7 | 2
  Week 100 | 0.99 (0.445) | 1.00 (0.424)
  Week 112: number analyzed (Participants) | 5 | 2
  Week 112 | 1.26 (0.508) | 1.10 (0.283)

15. Secondary Outcome: Change From Baseline in Mean Post-Baseline Serum Phosphorus Level to Week 64
Description: The ANCOVA model includes change in serum phosphorus from baseline to mean post-baseline as the dependent variable, treatment group, baseline age and baseline RSS stratification as factors, baseline phosphorous measure as a covariate.
Time Frame: Baseline, Weeks 1, 4, 8, 16, 24, 32, 40, 52, 64
Population: PD Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
mg/dL | 0.24 (0.058) | 0.98 (0.061)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Test type: Superiority; p < 0.0001, ANCOVA; difference in LS means = 0.74, 95% CI 2-sided [0.58 to 0.91] — Difference (KRN23 - Oral Phosphate/Active Vitamin D)

16. Secondary Outcome: Change From Baseline in Mean Post-Baseline Serum Phosphorus Level to Week 140 (During Treatment With Burosumab)
Time Frame: Burosumab arm: Baseline, Week 1, 4, 8, 16, 24, 32, 40, 52, 64, 66, 68, 76, 88, 100, 112, 124, 140; Active Control arm: Baseline, Week 68, 76, 88, 100, 112, 124, 140
Population: PD Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 26 | 29
mg/dL | 1.05 (0.310) | 0.93 (0.336)

17. Secondary Outcome: Percentage of Participants Reaching the Normal Range of Serum Phosphorus Concentration (3.2 - 6.1 mg/dL)
Time Frame: Burosumab arm: Baseline, up to Week 140; Active Control arm: Baseline, Week 68 up to Week 140
Population: PD Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data.
Measure: Number; unit: percentage of participants
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
percentage of participants | 75.0 | 96.6

18. Secondary Outcome: Change From Baseline Over Time in 1,25-Dihydroxyvitamin D, up to Week 64
Description: The GEE model includes change from baseline for 1, 25-Dihydroxyvitamin D measurement as the dependent variable, treatment group, visit, interaction between treatment group by visit, baseline age and baseline RSS stratification as factors, baseline 1, 25-Dihydroxyvitamin D measure as a covariate, with exchangeable covariance structure. The GEE model included data up to Week 64.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16, 24, 32, 33, 40, 52, 64
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 30 | 28
pg/mL
  Week 1: number analyzed (Participants) | 29 | 27
  Week 1 | 19.81 (2.758) | 68.09 (5.251)
  Week 2: number analyzed (Participants) | 0 | 24
  Week 2 |  | 31.78 (5.130)
  Week 4: number analyzed (Participants) | 30 | 27
  Week 4 | 12.77 (2.998) | 33.86 (3.561)
  Week 8 | 15.10 (2.528) | 30.85 (3.830)
  Week 12: number analyzed (Participants) | 0 | 24
  Week 12 |  | 33.43 (3.176)
  Week 16: number analyzed (Participants) | 27 | 28
  Week 16 | 19.41 (3.757) | 32.38 (3.032)
  Week 24: number analyzed (Participants) | 28 | 27
  Week 24 | 17.46 (2.905) | 28.35 (3.113)
  Week 32: number analyzed (Participants) | 29 | 28
  Week 32 | 17.25 (3.156) | 23.49 (2.439)
  Week 33: number analyzed (Participants) | 0 | 24
  Week 33 |  | 31.50 (3.423)
  Week 40: number analyzed (Participants) | 27 | 25
  Week 40 | 18.42 (3.594) | 29.63 (3.721)
  Week 52: number analyzed (Participants) | 29 | 27
  Week 52 | 8.74 (3.866) | 13.75 (2.862)
  Week 64: number analyzed (Participants) | 29 | 27
  Week 64 | 1.19 (2.785) | 9.89 (2.235)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Week 1; Test type: Superiority; p < 0.0001, GEE model; difference = 48.27, 95% CI 2-sided [36.53 to 60.02] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 2: Comparison: Active Control vs Burosumab; Week 4; Test type: Superiority; p < 0.0001, GEE model; difference = 21.09, 95% CI 2-sided [12.01 to 30.16] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 3: Comparison: Active Control vs Burosumab; Week 8; Test type: Superiority; p = 0.0010, GEE model; difference = 15.75, 95% CI 2-sided [6.35 to 25.15] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 4: Comparison: Active Control vs Burosumab; Week 16; Test type: Superiority; p = 0.0078, GEE model; difference = 12.97, 95% CI 2-sided [3.41 to 22.53] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 5: Comparison: Active Control vs Burosumab; Week 24; Test type: Superiority; p = 0.0101, GEE model; difference = 10.89, 95% CI 2-sided [2.59 to 19.19] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 6: Comparison: Active Control vs Burosumab; Week 32; Test type: Superiority; p = 0.1165, GEE model; difference = 6.23, 95% CI 2-sided [-1.55 to 14.02] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 7: Comparison: Active Control vs Burosumab; Week 40; Test type: Superiority; p = 0.0317, GEE model; difference = 11.21, 95% CI 2-sided [0.98 to 21.44] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 8: Comparison: Active Control vs Burosumab; Week 52; Test type: Superiority; p = 0.3044, GEE model; difference = 5.01, 95% CI 2-sided [-4.55 to 14.56] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 9: Comparison: Active Control vs Burosumab; Week 64; Test type: Superiority; p = 0.0145, GEE model; difference = 8.70, 95% CI 2-sided [1.72 to 15.68] — Difference (Burosumab - Oral Phosphate/Active Vitamin D

19. Secondary Outcome: Change From Baseline Over Time in 1,25-Dihydroxyvitamin D, Weeks 68 to 112
Time Frame: Baseline, Weeks 68, 76, 88, 100, 112
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 25 | 21
pg/mL
  Week 68: number analyzed (Participants) | 25 | 1
  Week 68 | 22.12 (23.950) | -9.80 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 21 | 21
  Week 76 | 19.05 (22.612) | 12.80 (20.093)
  Week 88: number analyzed (Participants) | 14 | 10
  Week 88 | 24.58 (17.787) | 11.76 (22.874)
  Week 100: number analyzed (Participants) | 6 | 2
  Week 100 | 33.57 (16.591) | 13.25 (1.061)
  Week 112: number analyzed (Participants) | 5 | 2
  Week 112 | 29.94 (15.402) | 31.05 (33.729)

20. Secondary Outcome: Change From Baseline Over Time in TmP/GFR, up to Week 64
Description: Serum phosphorus and TRP measurements were used in the calculation of TmP/GFR.
  The GEE model includes change from baseline for TmP/GFR measurement as the dependent variable, treatment group, visit, interaction between treatment group by visit, baseline age and baseline RSS stratification as factors, baseline TmP/GFR measure as a covariate, with exchangeable covariance structure. The GEE model included data up to Week 64.
Time Frame: Baseline, Weeks 4, 8, 16, 24, 32, 40, 52, 64
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 30 | 24
mg/dL
  Week 4: number analyzed (Participants) | 28 | 23
  Week 4 | -0.17 (0.065) | 1.48 (0.173)
  Week 8: number analyzed (Participants) | 27 | 24
  Week 8 | -0.20 (0.057) | 1.22 (0.101)
  Week 16: number analyzed (Participants) | 26 | 24
  Week 16 | -0.15 (0.085) | 1.00 (0.139)
  Week 24: number analyzed (Participants) | 29 | 23
  Week 24 | -0.12 (0.072) | 0.99 (0.134)
  Week 32: number analyzed (Participants) | 29 | 22
  Week 32 | -0.10 (0.062) | 1.14 (0.115)
  Week 40: number analyzed (Participants) | 28 | 23
  Week 40 | -0.15 (0.053) | 1.20 (0.113)
  Week 52: number analyzed (Participants) | 28 | 22
  Week 52 | -0.12 (0.069) | 1.13 (0.124)
  Week 64: number analyzed (Participants) | 30 | 23
  Week 64 | -0.09 (0.070) | 1.16 (0.127)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Week 4; Test type: Superiority; p < 0.0001, GEE model; difference = 1.65, 95% CI 2-sided [1.28 to 2.02] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 2: Comparison: Active Control vs Burosumab; Week 8; Test type: Superiority; p < 0.0001, GEE model; difference = 1.42, 95% CI 2-sided [1.19 to 1.64] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 3: Comparison: Active Control vs Burosumab; Week 16; Test type: Superiority; p < 0.0001, GEE model; difference = 1.16, 95% CI 2-sided [0.84 to 1.48]
Statistical Analysis 4: Comparison: Active Control vs Burosumab; Week 24; Test type: Superiority; p < 0.0001, GEE model; difference = 1.11, 95% CI 2-sided [0.80 to 1.41] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 5: Comparison: Active Control vs Burosumab; Week 32; Test type: Superiority; p < 0.0001, GEE model; difference = 1.24, 95% CI 2-sided [0.98 to 1.51]
Statistical Analysis 6: Comparison: Active Control vs Burosumab; Week 40; Test type: Superiority; p < 0.0001, GEE model; difference = 1.35, 95% CI 2-sided [1.10 to 1.60] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 7: Comparison: Active Control vs Burosumab; Week 52; Test type: Superiority; p < 0.0001, GEE model; difference = 1.26, 95% CI 2-sided [0.97 to 1.54] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 8: Comparison: Active Control vs Burosumab; Week 64; Test type: Superiority; p < 0.0001, GEE model; difference = 1.25, 95% CI 2-sided [0.96 to 1.54] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)

21. Secondary Outcome: Change From Baseline Over Time in TmP/GFR, Week 68 to 112
Description: Serum phosphorus and TRP measurements were used in the calculation of TmP/GFR.
Time Frame: Baseline, Weeks 68, 76, 88, 112
Population: PD Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data. Participants with data at given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 24 | 7
mg/dL
  Week 68: number analyzed (Participants) | 24 | 1
  Week 68 | 1.61 (0.705) | 1.65 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 4 | 4
  Week 76 | 1.18 (0.758) | 0.59 (0.429)
  Week 88: number analyzed (Participants) | 14 | 7
  Week 88 | 1.33 (0.480) | 0.95 (0.620)
  Week 112: number analyzed (Participants) | 3 | 2
  Week 112 | 1.56 (0.233) | 1.32 (0.233)

22. Secondary Outcome: Change From Baseline Over Time in Serum ALP, up to Week 64
Description: The GEE model includes change from baseline for ALP measurement as the dependent variable, treatment group, visit, interaction between treatment group by visit, baseline age and baseline RSS stratification as factors, baseline ALP measure as a covariate, with exchangeable covariance structure. The GEE model included data up to Week 64.
Time Frame: Baseline, Weeks 16, 24, 40, 52, 64
Population: PD Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
U/L
  Week 16 | -5.43 (17.885) | -97.97 (11.281)
  Week 24 | -22.43 (15.074) | -108.00 (16.225)
  Week 40 | -34.78 (18.132) | -130.72 (12.365)
  Week 52 | -50.03 (18.641) | -161.31 (11.674)
  Week 64 | -28.06 (19.980) | -174.62 (13.427)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Week 16; Test type: Superiority; p < 0.0001, GEE model; difference = -92.53, 95% CI 2-sided [-131.40 to -53.66] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 2: Comparison: Active Control vs Burosumab; Week 24; Test type: Superiority; p < 0.0001, GEE model; difference = -85.57, 95% CI 2-sided [-126.37 to -44.76] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 3: Comparison: Active Control vs Burosumab; Week 40; Test type: Superiority; p < 0.0001, GEE model; difference = -95.95, 95% CI 2-sided [-136.05 to -55.84] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 4: Comparison: Active Control vs Burosumab; Week 52; Test type: Superiority; p < 0.0001, GEE model; difference = -111.28, 95% CI 2-sided [-152.08 to -70.49] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)
Statistical Analysis 5: Comparison: Active Control vs Burosumab; Week 64; Test type: Superiority; p < 0.0001, GEE model; difference = -146.56, 95% CI 2-sided [-191.61 to -101.52] — Difference (Burosumab - Oral Phosphate/Active Vitamin D)

23. Secondary Outcome: Change From Baseline Over Time in Serum ALP, Week 68 to 112
Time Frame: Baseline, Weeks 68, 76, 88, 100, 112
Population: PD Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 26 | 22
U/L
  Week 68: number analyzed (Participants) | 26 | 1
  Week 68 | -82.73 (83.683) | -184.00 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 22 | 22
  Week 76 | -106.73 (73.316) | -166.73 (87.700)
  Week 88: number analyzed (Participants) | 16 | 11
  Week 88 | -146.56 (73.120) | -154.55 (48.148)
  Week 100: number analyzed (Participants) | 7 | 2
  Week 100 | -83.14 (104.675) | -184.00 (48.083)
  Week 112: number analyzed (Participants) | 5 | 2
  Week 112 | -104.80 (80.350) | -172.00 (26.870)

24. Secondary Outcome: Percent Change From Baseline Over Time in Serum ALP, up to Week 112
Description: Decreases indicate improvement.
Time Frame: Baseline, Weeks 16, 24, 40, 52, 64, 68, 76, 88, 100, 112
Population: PD Analysis Set: all participants who received at least one dose of study therapy and had evaluable serum data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 32 | 29
percent change
  Week 16: number analyzed (Participants) | 29 | 29
  Week 16 | 0.41 (21.021) | -18.39 (10.815)
  Week 24 | -3.21 (15.827) | -19.88 (17.642)
  Week 40 | -6.85 (16.493) | -24.38 (13.498)
  Week 52 | -8.60 (19.027) | -30.60 (11.852)
  Week 64 | -4.60 (20.711) | -32.78 (13.095)
  Week 68: number analyzed (Participants) | 26 | 1
  Week 68 | -14.66 (14.760) | -38.02 (NA) — 1 participant analyzed
  Week 76: number analyzed (Participants) | 22 | 22
  Week 76 | -20.49 (13.926) | -31.42 (13.422)
  Week 88: number analyzed (Participants) | 16 | 11
  Week 88 | -28.77 (12.201) | -32.02 (10.610)
  Week 100: number analyzed (Participants) | 7 | 2
  Week 100 | -16.06 (23.703) | -39.29 (11.460)
  Week 112: number analyzed (Participants) | 5 | 2
  Week 112 | -21.00 (15.053) | -36.67 (6.868)

25. Secondary Outcome: Change From Baseline in the PROMIS Pediatric Pain Interference, Physical Function Mobility and Fatigue Domain Scores (For Participants ≥ 5 Years of Age at the Screening Visit) at Week 40
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013), (NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Pain Interference Domain, decreases indicate less pain, for the Physical Function Mobility Domain, increases indicate greater mobility and for the Fatigue Domain, decreases indicate less fatigue.
Time Frame: Baseline, Week 40
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 20 | 15
T-score
  Pain Interference Domain Score | -0.29 (1.539) | -5.31 (1.705)
  Physical Function Mobility Domain Score | 0.10 (0.966) | 2.78 (1.336)
  Fatigue Domain Score | -1.05 (1.754) | -4.29 (1.709)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; Pain Interference Domain. 2-sided p value per GEE model, which included change from baseline for the parameter as the dependent variable, treatment group, visit, interaction between treatment group by visit, baseline age and baseline RSS stratification as factors, baseline parameter measure as a covariate, with exchangeable covariance structure; Test type: Superiority; p = 0.0212, GEE model; difference in LS means = -5.02, 95% CI 2-sided [-9.29 to -0.75]
Statistical Analysis 2: Comparison: Active Control vs Burosumab; Physical Function Mobility Domain. 2-sided p value per GEE model, which included change from baseline for the parameter as the dependent variable, treatment group, visit, interaction between treatment group by visit, baseline age and baseline RSS stratification as factors, baseline parameter measure as a covariate, with exchangeable covariance structure; Test type: Superiority; p = 0.1009, GEE model; difference in LS means = 2.68, 95% CI 2-sided [-0.52 to 5.89]
Statistical Analysis 3: Comparison: Active Control vs Burosumab; Fatigue Domain. 2-sided p value per GEE model, which included change from baseline for the parameter as the dependent variable, treatment group, visit, interaction between treatment group by visit, baseline age and baseline RSS stratification as factors, baseline parameter measure as a covariate, with exchangeable covariance structure; Test type: Superiority; p = 0.1676, GEE model; difference in LS means = -3.25, 95% CI 2-sided [-7.86 to 1.37]

26. Secondary Outcome: Change From Baseline in the PROMIS Pediatric Pain Interference, Physical Function Mobility and Fatigue Domain Scores (For Participants ≥ 5 Years of Age at the Screening Visit) at Week 64
Description: as for outcome 25
Time Frame: Baseline, Week 64
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 20 | 15
T-score
  Pain Interference Domain Score | -1.29 (1.267) | -3.55 (1.873)
  Physical Function Mobility Domain Score | 0.92 (0.962) | 2.82 (1.648)
  Fatigue Domain Score | -2.57 (1.547) | -3.65 (2.119)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.3091, GEE model; difference in LS means = -2.26, 95% CI 2-sided [-6.61 to 2.09]
Statistical Analysis 2: Comparison: Active Control vs Burosumab; [analysis description as in outcome 25, analysis 2]; Test type: Superiority; p = 0.3145, GEE model; difference in LS means = 1.90, 95% CI 2-sided [-1.80 to 5.59]
Statistical Analysis 3: Comparison: Active Control vs Burosumab; [analysis description as in outcome 25, analysis 3]; Test type: Superiority; p = 0.6810, GEE model; difference in LS means = -1.08, 95% CI 2-sided [-6.21 to 4.06]

27. Secondary Outcome: Change From Baseline in the FPS-R (For Participants ≥ 5 Years of Age at the Screening Visit) at Week 40
Description: The FPS-R is a dimensionless 10 point Likert scale used to assess self-reported pain intensity on a scale from 0 (no pain) to 10 (most pain you can imagine). Greater pain scores are indicative of more severe pain.
Time Frame: Baseline, Week 40
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 20 | 15
units on a scale | 0.02 (0.323) | 0.03 (0.323)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; GEE model includes change from baseline for FPS-R as the dependent variable, treatment group, visit, interaction between treatment group by visit and baseline RSS stratification as factors, baseline FPS-R as a covariate, with exchangeable covariance structure. The LS Mean, SE, 95% CI and 2-sided p-value are from the GEE model; Test type: Superiority; p = 0.9862, GEE model; Difference in LS Means = 0.01, 95% CI 2-sided [-0.79 to 0.80]

28. Secondary Outcome: Change From Baseline in the FPS-R (For Participants ≥ 5 Years of Age at the Screening Visit) at Week 64
Description: as for outcome 27
Time Frame: Baseline, Week 64
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 19 | 15
units on a scale | 0.04 (0.270) | -0.01 (0.234)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p = 0.8786, GEE model; difference in LS means = 0.05, 95% CI 2-sided [-0.58 to 0.68]

29. Secondary Outcome: Change From Baseline in the 6MWT Total Distance at Week 40
Description: The total distance walked (meters) in a 6-minute period was measured in participants ≥ 5 years of age at the Screening Visit who were able to complete the test.
Time Frame: Baseline, Week 40
Population: Full Analysis Set: all randomized participants who received at least one dose of assigned medication and had at least one post-baseline assessment. Participants with an assessment at Week 40 in subjects ≥ 5 years who were able to complete the test.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 20 | 13
meters | 3.65 (14.060) | 47.10 (15.768)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; 2-sided p value per GEE model, which included change from baseline for the parameter as the dependent variable, treatment group, visit, interaction between treatment group by visit, baseline age and baseline RSS stratification as factors, baseline parameter measure as a covariate, with exchangeable covariance structure; Test type: Superiority; p = 0.0514, GEE model; difference in LS means = 43.46, 95% CI 2-sided [-0.26 to 87.17]

30. Secondary Outcome: Change From Baseline in the 6MWT Total Distance at Week 64
Description: as for outcome 29
Time Frame: Baseline, Week 64
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 20 | 13
meters | 29.28 (16.834) | 74.83 (12.513)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0399, GEE model; difference in LS means = 45.55, 95% CI 2-sided [2.09 to 89.02]

31. Secondary Outcome: Percent of Predicted Normal in the 6MWT Total Distance at Week 40
Description: The total distance walked (meters) in a 6-minute period was measured in participants ≥ 5 years of age at the Screening Visit who were able to complete the test, and the percent predicted distance based on normative data for age and gender was estimated.
Time Frame: Baseline, Week 40
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percent of predicted meters
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 20 | 13
percent of predicted meters | -1.14 (2.224) | 5.59 (2.633)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0633, GEE model; difference in LS means = 6.72, 95% CI 2-sided [-0.37 to 13.82]

32. Secondary Outcome: Percent of Predicted Normal in the 6MWT Total Distance at Week 64
Description: as for outcome 31
Time Frame: Baseline, Week 64
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: percent of predicted meters
Arm/Group | Active Control | Burosumab
Number analyzed (Participants) | 20 | 13
percent of predicted meters | 1.88 (2.789) | 9.15 (2.056)
Statistical Analysis 1: Comparison: Active Control vs Burosumab; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0496, GEE model; difference in LS means = 7.27, 95% CI 2-sided [0.01 to 14.52]

ADVERSE EVENTS:
Time Frame: Up to Week 64 in the Treatment Period and up to Week 140 in the Long Term Extension Period, plus up to 12 weeks ±1 week after the last dose of study drug.
Groups:
- Oral Phosphate/Active Vitamin D (Treatment Period): Multiple daily doses of oral phosphate and one or more daily doses of active vitamin D therapy, titrated and individualized by the investigator based on published recommendations during the Treatment Period (up to Week 64).
- Burosumab (Treatment Period): Burosumab 0.8 mg/kg starting dose, administered Q2W by SC injection during the Treatment Period (up to Week 64).
- Oral Phosphate/Active Vitamin D->Burosumab (Extension Period): Multiple daily doses of oral phosphate and one or more daily doses of active vitamin D therapy, titrated and individualized by the investigator based on published recommendations during the Treatment Period (up to Week 64). During the Treatment Extension Period (Week 64 to Week 140), participants crossed over to receive a starting dose of SC burosumab 0.8 mg/kg Q2W. Participants in Japan and Korea did not enter the Treatment Extension Period.
- Burosumab->Burosumab (Treatment Period and Extension Period): Burosumab 0.8 mg/kg starting dose, administered Q2W by SC injection during the Treatment Period (up to Week 64). During the Treatment Extension Period (Week 64 to Week 140), participants continued to receive a starting dose of SC burosumab 0.8 mg/kg Q2W. Participants in Japan and Korea did not enter the Treatment Extension Period.
- Total Burosumab (Treatment Period and Extension Period): Burosumab 0.8 mg/kg starting dose, administered Q2W by SC injection at any time during the study.
Arm/Group | Oral Phosphate/Active Vitamin D (Treatment Period) | Burosumab (Treatment Period) | Oral Phosphate/Active Vitamin D->Burosumab (Extension Period) | Burosumab->Burosumab (Treatment Period and Extension Period) | Total Burosumab (Treatment Period and Extension Period)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29 | 0/26 | 0/29 | 0/55
Serious Adverse Events (participants affected / at risk) | 3/32 | 3/29 | 0/26 | 4/29 | 4/55
Other Adverse Events (participants affected / at risk) | 23/32 | 21/29 | 9/26 | 25/29 | 34/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Phosphate/Active Vitamin D (Treatment Period) (N=32) | Burosumab (Treatment Period) (N=29) | Oral Phosphate/Active Vitamin D->Burosumab (Extension Period) (N=26) | Burosumab->Burosumab (Treatment Period and Extension Period) (N=29) | Total Burosumab (Treatment Period and Extension Period) (N=55)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 1 | 1
Papilloedema (Eye disorders) | 0 | 0 | 0 | 1 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Phosphate/Active Vitamin D (Treatment Period) (N=32) | Burosumab (Treatment Period) (N=29) | Oral Phosphate/Active Vitamin D->Burosumab (Extension Period) (N=26) | Burosumab->Burosumab (Treatment Period and Extension Period) (N=29) | Total Burosumab (Treatment Period and Extension Period) (N=55)
Tooth Hypoplasia (Congenital, familial and genetic disorders) | 0 | 2 | 0 | 2 | 2
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 2
Ear Pain (Ear and labyrinth disorders) | 1 | 4 | 2 | 4 | 6
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 3 | 2 | 4 | 6
Constipation (Gastrointestinal disorders) | 0 | 5 | 2 | 5 | 7
Dental Caries (Gastrointestinal disorders) | 2 | 9 | 0 | 10 | 10
Diarrhoea (Gastrointestinal disorders) | 2 | 7 | 1 | 7 | 8
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 5 | 7
Teething (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 3
Tooth Loss (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3
Toothache (Gastrointestinal disorders) | 1 | 4 | 1 | 5 | 6
Vomiting (Gastrointestinal disorders) | 8 | 12 | 5 | 14 | 19
Fatigue (General disorders) | 2 | 1 | 1 | 2 | 3
Injection Site Bruising (General disorders) | 0 | 0 | 2 | 1 | 3
Injection Site Erosion (General disorders) | 0 | 2 | 0 | 2 | 2
Injection Site Erythema (General disorders) | 0 | 9 | 6 | 9 | 15
Injection Site Pruritus (General disorders) | 0 | 3 | 2 | 3 | 5
Injection Site Rash (General disorders) | 0 | 3 | 0 | 3 | 3
Injection Site Reaction (General disorders) | 0 | 7 | 2 | 8 | 10
Injection Site Swelling (General disorders) | 0 | 3 | 1 | 3 | 4
Injection Site Urticaria (General disorders) | 0 | 2 | 0 | 2 | 2
Pain (General disorders) | 0 | 2 | 0 | 3 | 3
Pyrexia (General disorders) | 7 | 16 | 7 | 17 | 24
Hypersensitivity (Immune system disorders) | 2 | 1 | 0 | 1 | 1
Seasonal Allergy (Immune system disorders) | 2 | 4 | 1 | 4 | 5
Ear Infection (Infections and infestations) | 3 | 2 | 1 | 3 | 4
Gastroenteritis (Infections and infestations) | 3 | 2 | 0 | 2 | 2
Gastroenteritis Viral (Infections and infestations) | 3 | 2 | 0 | 2 | 2
Influenza (Infections and infestations) | 6 | 4 | 0 | 4 | 4
Nasopharyngitis (Infections and infestations) | 14 | 11 | 6 | 15 | 21
Otitis Externa (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 4 | 2 | 0 | 3 | 3
Pharyngitis Streptococcal (Infections and infestations) | 1 | 1 | 1 | 2 | 3
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 2 | 2
Rhinitis (Infections and infestations) | 2 | 2 | 0 | 2 | 2
Tooth Abscess (Infections and infestations) | 3 | 8 | 2 | 9 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 3 | 0 | 3 | 3
Varicella (Infections and infestations) | 0 | 2 | 1 | 2 | 3
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 4 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 3 | 3
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2 | 2
Vitamin D Decreased (Investigations) | 1 | 6 | 1 | 6 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 5 | 0 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 13 | 3 | 13 | 16
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 2 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 | 11 | 3 | 11 | 14
Headache (Nervous system disorders) | 6 | 10 | 3 | 10 | 13
Migraine (Nervous system disorders) | 2 | 1 | 1 | 1 | 2
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 0 | 0 | 0 | 2 | 2
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 15 | 4 | 15 | 19
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 7 | 8
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3 | 6 | 9
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 3 | 8 | 11
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 4 | 4
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT02915705/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT02915705/SAP_001.pdf